CLINICAL TRIAL: NCT04385914
Title: Demographics and Outcomes of Pregnant COVID 19 Positive Women in a Community Health System
Brief Title: Demographics and Outcomes of COVID 19 in Pregnancy at a Community Based Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Farah Benarba, DO, Atlantic Health System
Other Study IDs: 1595116-1
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID positive patients
  Interventions: Other: COVID positive via testing
- COVID negative patients
  Interventions: Other: COVID positive via testing

INTERVENTIONS:
Other: COVID positive via testing — Following pregnancy outcomes whether they are COVID positive or negative

SUMMARY:
Demographics of pregnant COVID persons under investigation and those who were positive from March-May 2020. Looking at demographics including age, socio-economic status and pregnancy outcomes in these groups.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant, considered PUI or know COVID positive patient during pregnancy, and documentation of COVID symptoms within AHS.

Exclusion Criteria:

* Not pregnant, No documentation of COVID-19 symptoms within AHS.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: Pregnant patients who presented to AHS within March-May 2020
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Outcome | through study completion, approximately 1 year
  increased risk of preterm birth, preeclampsia, etc.

IPD SHARING:
Plan to Share IPD: No